CLINICAL TRIAL: NCT02009553
Title: Pre-procedural Information Sheet Reduces Anxiety of Patients Before Urodynamic Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 167/13; 167/13 (Other: Assaf Harofe Medical Center)
Record Dates: First submitted 2013-12-02; First posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Anxiety
Keywords: Anxiety; Urodynamics
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Information sheet, Applied: In this group, all patients will receive the information sheet one month before the procedure
  Interventions: Other: Information sheet
- Information sheet, not applied: In this group, patients will not receive a pre-procedural information sheet
  Interventions: Other: No information sheet

INTERVENTIONS:
Other: Information sheet
  Groups: Information sheet, Applied
Other: No information sheet
  Groups: Information sheet, not applied

SUMMARY:
Urodynamic study may lead to significant anxiety. Our hypothesis is that Urodynamic study is that pre-procedural explanation note about the test may reduce the anxiety level of the patients.

DETAILED DESCRIPTION:
Urodynamic study is one of the most common procedures in urological outpatient practice. Patients who wait for the tests may experience significant anxiety.

in this study, patients who are designated to have multichannel Urodynamic study will be randomized to two groups: group 1 - patients who received an explanation note about the test; group 2 - patients who did not receive the note. The explanation notes will be sent to the patients in group 1 by mail one month before the test.

Investigators will use the State Anxiety Inventory (SAI) in order to assess emotional distress immediately before the test. Comparison opf the anxiety level between the two groups will be performed.

ELIGIBILITY:
Inclusion Criteria:

All patients who will be referred for Urodynamic studies in order to evaluate lower urinary tract symptoms.

Exclusion Criteria:

1. inability to complete the questionnaire due to mental disorders
2. patients who had undergone Urodynamic study previously

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be designated to have multichannel Uridynamic study in our center.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Inventory | 10 minutes before the test
  Investigators will use the State Anxiety Inventory (SAI) in order to assess emotional distress. The SAI is a validated questionnaire composed of 20-items measures of anxiety (e.g. ''I am anxious''). Respondents will be requested to rate their endorsement of each item on a four-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Beer Yaakov, Zeriffin, Israel